CLINICAL TRIAL: NCT04671043
Title: Does Combined Caffeine and Carbohydrate Ingestion Counter the Exercise-mediated Fall in Glycaemia in Individuals With Type 1 Diabetes on Insulin Degludec? The DE-CAF Study
Brief Title: Caffeine Ingestion to Counter the Exercise-mediated Fall in Glycaemia in Type 1 Diabetes
Acronym: DE-CAF
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Insel Gruppe AG, University Hospital Bern (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Prevention
Other Study IDs: DE-CAF
Record Dates: First submitted 2020-12-10; First posted 2020-12-17 (Actual); Last update posted 2023-03-14 (Actual); Status verified 2023-03

CONDITIONS: Caffeine and Carbohydrate; Carbohydrate Only; Placebo
Keywords: caffeine; type 1 diabetes; exercise; hypoglycemia; glucose
MeSH Terms: conditions — Diabetes Mellitus, Type 1; Motor Activity; Hypoglycemia | interventions — Caffeine; Glucose

STUDY DESIGN:
Intervention Model Description: Single-centre, randomised, double-blind crossover design
Who Masked: Participant, Investigator
Masking Description: In each of the conditions, participants will receive a taste-matched drink containing either • caffeine and 10 g rapid-acting carbohydrate (CAF+lowCHO); 20 g rapid acting carbohydrate (20g CHO); or placebo. The drink will be made by an independent member of the research team to ensure that neither the investigators or participants know the order of the drinks (double-blind)
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- CAF+lowCHO (Experimental): A drink containing caffeine and 10 g rapid-acting carbohydrate (glucose) dissolved in 200 mL of tap water
  Interventions: Dietary Supplement: Caffeine and glucose
- 10g CHO (Active Comparator): A drink containing 10 g rapid-acting carbohydrate (glucose) dissolved in 200 mL of tap water
  Interventions: Dietary Supplement: Glucose alone
- placebo (Placebo Comparator): A drink containing an artificial sweetener (aspartame) dissolved in 200 mL of tap water
  Interventions: Dietary Supplement: Placebo

INTERVENTIONS:
Dietary Supplement: Caffeine and glucose — Caffeine and glucose powder dissolved in water
  Arms: CAF+lowCHO
Dietary Supplement: Glucose alone — Glucose powder dissolved in water
  Arms: 10g CHO
Dietary Supplement: Placebo — Artificial sweetener dissolved in water
  Arms: placebo

SUMMARY:
This project will aim to investigate the clinical efficacy and metabolic effects of a pre-exercise dose of caffeine with a low (10g) dose of carbohydrate (CAF+lowCHO) without modification of insulin degludec on exercise metabolism in people with T1D.

DETAILED DESCRIPTION:
Treatment of type 1 diabetes (T1D) involves lifelong use of exogenous insulin to manage blood glucose concentration. As with the rest of the population, people living with T1D are recommended to engage in regular exercise for a variety of health and fitness reasons . However, glycaemic control during exercise remains a particular challenge for this population due to rapid changes in insulin sensitivity and the impact of additional hormones which increase the risk of exercise-related hypoglycaemia. Current guidelines to prevent exercise-induced hypoglycaemia suggest insulin dose reduction and/or ingestion of carbohydrates in the context of the exercise bout. However, these adaptations are often difficult to apply, as insulin dose adjustments require knowledge of insulin pharmacokinetics and advanced planning which is not always possible. None of these strategies provide complete assurance that hypoglycaemia will not occur and high carbohydrate intake can be counterproductive if weight management is the target. Furthermore, modern very long-acting insulin analogues, which are favoured by many people with T1D, do not offer the option to rapidly or transiently reduce insulin before exercise. When using such insulins, dose reductions may take two to three days to achieve an adapted steady state, increasing the risk of inadequate insulin following exercise. Collectively, these factors increase the risk of further deterring patients from exercise. Simple, alternative strategies to reduce the risk of hypoglycaemia, both during and after exercise are needed.

Caffeine (1,3,7-trimethylxanthine) is the most commonly consumed chemical stimulant in the world that is naturally found in many foods and is frequently added to sports supplements due to its ergogenic effects in a range of sporting events. Caffeine has numerous physiological effects throughout the body including increased lipolysis in adipose tissues and hepatic glucose production in the liver alongside a decrease in glucose uptake in skeletal muscle. These responses have led to the suggestion that acute caffeine intake may attenuate exercise-associated hypoglycaemia in people with T1D. Ingestion of modest amounts of caffeine (200-250 mg, equivalent to 3-4 cups of coffee each day) has been shown to augment the symptomatic and hormonal responses to hypoglycaemia in participants with and without T1D. Caffeine has also been shown to reduce the frequency of moderate episodes of hypoglycaemia occurring overnight. The paucity of data on caffeine and exercise in individuals with T1D, in conjunction with caffeine's popularity both socially and as a sports supplement, suggests this deserves further attention.

A clear example whereby caffeine supplementation may be of use is in patients using an ultra-long acting basal insulin analogue such as insulin degludec. The administration is via subcutaneous injection once daily, and it has a duration of action that lasts up to 42 hours (compared to 18 to 26 hours provided by other marketed long-acting insulins such as insulin glargine and insulin detemir). On average, the half-life at steady state is approximately 25 hours independent of dose. Compared to the other basal insulin analogues, the risk of hypoglycaemia appears to be lower with insulin degludec, however, hypoglycaemia still occurs. In the case of physical exercise, the inability of the patient using such long-acting insulins to make rapid adjustments can translate to the occurrence of exercise-related hypoglycaemia due to an inability to reduce insulin already onboard, hence the need for new strategies to prevent this undesired phenomenon. When using such insulins, dose reductions may take two to three days to achieve an adapted steady state, increasing the risk of inadequate insulin following exercise. Applying a novel in-house developed lipid chromatography-mass spectrometry (LC-MS) assay, members of our research group observed that a single bout of aerobic exercise increases systemic insulin degludec concentrations in adults on stable basal insulin degludec regimens. Therefore, if these individuals wish to engage in regular exercise, as recommended in international guidelines, current treatment strategies may not be sufficient. For patients treated with modern basal insulin analogues, it seems more adequate not to modify the ultra-long acting insulin doses, as this can often result in more confusion than improvement, but to apply alternative strategies for recreational exercise. Caffeine ingestion pre or post exercise may offer a simple means to better manage glycaemia in the context of exercise in patients using these insulins and have the added benefit of reducing carbohydrate requirements in the context of exercise.

ELIGIBILITY:
Inclusion Criteria:

* Type 1 diabetes for ≥1 year and negative C-peptide (<100pmol/l)
* Male and female aged 18-45 years old
* HbA1c <8.5% (69 mmol/mol) based on analysis from the central laboratory unit of Bern University Hospital
* Using multiple daily injections
* Using insulin degludec (Tresiba; Novo Nordisk A/S, Bagsværd, Denmark) as basal insulin for a minimum of 3 months
* Written informed consent
* Able and willing to adhere to safe contraception during the study and for 2 weeks after completion of the study. Safe contraception comprises double barrier methods (hormonal contraception [like: oral contraceptive pills or intrauterine contraceptive devices] together with a mechanical barrier [like: condom, diaphragm]).

Exclusion Criteria:

* Physical or psychological disease likely to interfere with the normal conduct of the study as judged by the investigator
* Continuous subcutaneous insulin infusion (using an insulin pump)
* Hypoglycaemic unawareness (Gold likert score ≥4) or having experienced any episode of a severe hypoglycaemic event within the last 6 months (i.e. need of third-party assistance).
* Current treatment with drugs known to interfere with metabolism e.g. systemic corticosteroids, SGLT2 inhibitors, Glucagon like 1 peptide- receptor agonists, or metformin.
* Relevant diabetic complications as judged by the investigator and based on medical record check (no cardiovascular disease and no significant microvascular disease)
* Microalbuminuria (as defined by area under the curve >30 mg/g)
* Body mass index more than or equal to 30 kg/m2
* Uncontrolled hypertension (>180/100 mmHg)
* Pregnant or planning to become pregnant during the study period (females only)
* Breastfeeding

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 21 (Actual)
Dates: Start 2022-02-04 (Actual); Primary Completion 2023-02-02 (Actual); Study Completion 2023-02-02 (Actual)

PRIMARY OUTCOMES:
Hypoglycaemia | 60 minutes from start of exercise
  Time to hypoglycaemia (plasma glucose <3.9mmol/l) during the 60 min of exercise

SECONDARY OUTCOMES:
Change in blood glucose concentration | 60 minutes from start of exercise
  Change in blood glucose concentration, calculated based on the participants' glucose at the start of exercise and the last value measured at the end of exercise. If the exercise is stopped early because of hypoglycaemia, the last exercise glucose value will be used for analysis.
Mean glucose concentration | 60 minutes from start of exercise
  Mean glucose concentration during the exercise bout
Area under the glucose curve | 60 minutes from start of exercise
  Area under the glucose curve during exercise
%-Time in target glycaemic range during recovery | 24 hours
  Time in target glycaemic range (4-10 mmol/l) in the recovery period and overnight
%-Time in target glycaemic range during exercise | 60 minutes
  Time in target glycaemic range (4-10 mmol/l) during exercise
Incidence of hypoglycaemia during exercise | 60 minutes
  Incidence of hypoglycaemia (≤3.9 mmol/l) during exercise
Incidence of hypoglycaemia during recovery | 24 hours
  Incidence of hypoglycaemia (≤3.9 mmol/l for 15 min or more) during the 24 hour post exercise recovery period
% Time below target range (< 3.9 mmol/L) during nighttime after exercise | 12:00 am until 06:00 am after each exercise visit
  The % time of glucose sensor measurements < 3.9 mmol/L in the night following the exercise visits will be documented
% Time below target range (> 10.0 mmol/L) during nighttime after exercise | 12:00 am until 06:00 am after each exercise visit
  The % time of glucose sensor measurements > 10.0 mmol/L in the night following the exercise visits will be documented
Mean sensor glucose overnight | 12:00 am until 06:00 am after each exercise visit
  The mean sensor glucose in mmol/L in the nights following the exercise visits will be documented
Area under the glucose curve post exercise | 30 minutes after stop of exercise
  The sensor glucose in mmol/L within 30 minutes following the exercise visits will be documented and the area under the curve will be calculated

CONTACTS AND LOCATIONS:
Overall Officials: Christoph Stettler, MD, Principal Investigator — University of Bern
Locations (1):
- Department of Diabetes, Endocrinology, Nutritional Medicine and Metabolism, Inselspital, Bern University Hospital and University of Bern, Bern, Switzerland, Bern, Switzerland

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Brazeau AS, Rabasa-Lhoret R, Strychar I, Mircescu H. Barriers to physical activity among patients with type 1 diabetes. Diabetes Care. 2008 Nov;31(11):2108-9. doi: 10.2337/dc08-0720. Epub 2008 Aug 8. PMID 18689694
- [Background] Buzzetti R, Zampetti S, Pozzilli P. Impact of obesity on the increasing incidence of type 1 diabetes. Diabetes Obes Metab. 2020 Jul;22(7):1009-1013. doi: 10.1111/dom.14022. Epub 2020 Mar 24. PMID 32157790
- [Background] Campbell MD, Walker M, Bracken RM, Turner D, Stevenson EJ, Gonzalez JT, Shaw JA, West DJ. Insulin therapy and dietary adjustments to normalize glycemia and prevent nocturnal hypoglycemia after evening exercise in type 1 diabetes: a randomized controlled trial. BMJ Open Diabetes Res Care. 2015 May 12;3(1):e000085. doi: 10.1136/bmjdrc-2015-000085. eCollection 2015. PMID 26019878
- [Background] Colberg SR, Sigal RJ, Yardley JE, Riddell MC, Dunstan DW, Dempsey PC, Horton ES, Castorino K, Tate DF. Physical Activity/Exercise and Diabetes: A Position Statement of the American Diabetes Association. Diabetes Care. 2016 Nov;39(11):2065-2079. doi: 10.2337/dc16-1728. No abstract available. PMID 27926890
- [Background] Costill DL, Dalsky GP, Fink WJ. Effects of caffeine ingestion on metabolism and exercise performance. Med Sci Sports. 1978 Fall;10(3):155-8. PMID 723503
- [Background] Debrah K, Sherwin RS, Murphy J, Kerr D. Effect of caffeine on recognition of and physiological responses to hypoglycaemia in insulin-dependent diabetes. Lancet. 1996 Jan 6;347(8993):19-24. doi: 10.1016/s0140-6736(96)91557-3. PMID 8531542
- [Background] Dedrick S, Sundaresh B, Huang Q, Brady C, Yoo T, Cronin C, Rudnicki C, Flood M, Momeni B, Ludvigsson J, Altindis E. The Role of Gut Microbiota and Environmental Factors in Type 1 Diabetes Pathogenesis. Front Endocrinol (Lausanne). 2020 Feb 26;11:78. doi: 10.3389/fendo.2020.00078. eCollection 2020. PMID 32174888
- [Background] Francescato MP, Geat M, Fusi S, Stupar G, Noacco C, Cattin L. Carbohydrate requirement and insulin concentration during moderate exercise in type 1 diabetic patients. Metabolism. 2004 Sep;53(9):1126-30. doi: 10.1016/j.metabol.2004.03.015. PMID 15334372
- [Background] Ganio MS, Klau JF, Casa DJ, Armstrong LE, Maresh CM. Effect of caffeine on sport-specific endurance performance: a systematic review. J Strength Cond Res. 2009 Jan;23(1):315-24. doi: 10.1519/JSC.0b013e31818b979a. PMID 19077738
- [Background] Graham TE, Sathasivam P, Rowland M, Marko N, Greer F, Battram D. Caffeine ingestion elevates plasma insulin response in humans during an oral glucose tolerance test. Can J Physiol Pharmacol. 2001 Jul;79(7):559-65. PMID 11478588
- [Background] Greer F, Hudson R, Ross R, Graham T. Caffeine ingestion decreases glucose disposal during a hyperinsulinemic-euglycemic clamp in sedentary humans. Diabetes. 2001 Oct;50(10):2349-54. doi: 10.2337/diabetes.50.10.2349. PMID 11574419
- [Background] Jackman M, Wendling P, Friars D, Graham TE. Metabolic catecholamine, and endurance responses to caffeine during intense exercise. J Appl Physiol (1985). 1996 Oct;81(4):1658-63. doi: 10.1152/jappl.1996.81.4.1658. PMID 8904583
- [Background] Kerr D, Sherwin RS, Pavalkis F, Fayad PB, Sikorski L, Rife F, Tamborlane WV, During MJ. Effect of caffeine on the recognition of and responses to hypoglycemia in humans. Ann Intern Med. 1993 Oct 15;119(8):799-804. doi: 10.7326/0003-4819-119-8-199310150-00005. PMID 8379601
- [Background] Kosinski C, Herzig D, Laesser CI, Nakas CT, Melmer A, Vogt A, Vogt B, Laimer M, Bally L, Stettler C. A Single Load of Fructose Attenuates the Risk of Exercise-Induced Hypoglycemia in Adults With Type 1 Diabetes on Ultra-Long-Acting Basal Insulin: A Randomized, Open-Label, Crossover Proof-of-Principle Study. Diabetes Care. 2020 Sep;43(9):2010-2016. doi: 10.2337/dc19-2250. Epub 2020 Jun 26. PMID 32591421
- [Background] Lane W, Bailey TS, Gerety G, Gumprecht J, Philis-Tsimikas A, Hansen CT, Nielsen TSS, Warren M; Group Information; SWITCH 1. Effect of Insulin Degludec vs Insulin Glargine U100 on Hypoglycemia in Patients With Type 1 Diabetes: The SWITCH 1 Randomized Clinical Trial. JAMA. 2017 Jul 4;318(1):33-44. doi: 10.1001/jama.2017.7115. PMID 28672316
- [Background] Lascar N, Kennedy A, Hancock B, Jenkins D, Andrews RC, Greenfield S, Narendran P. Attitudes and barriers to exercise in adults with type 1 diabetes (T1DM) and how best to address them: a qualitative study. PLoS One. 2014 Sep 19;9(9):e108019. doi: 10.1371/journal.pone.0108019. eCollection 2014. PMID 25237905
- [Background] Mayer-Davis EJ, Lawrence JM, Dabelea D, Divers J, Isom S, Dolan L, Imperatore G, Linder B, Marcovina S, Pettitt DJ, Pihoker C, Saydah S, Wagenknecht L; SEARCH for Diabetes in Youth Study. Incidence Trends of Type 1 and Type 2 Diabetes among Youths, 2002-2012. N Engl J Med. 2017 Apr 13;376(15):1419-1429. doi: 10.1056/NEJMoa1610187. PMID 28402773
- [Background] Richardson T, Thomas P, Ryder J, Kerr D. Influence of caffeine on frequency of hypoglycemia detected by continuous interstitial glucose monitoring system in patients with long-standing type 1 diabetes. Diabetes Care. 2005 Jun;28(6):1316-20. doi: 10.2337/diacare.28.6.1316. PMID 15920045
- [Background] Riddell MC, Gallen IW, Smart CE, Taplin CE, Adolfsson P, Lumb AN, Kowalski A, Rabasa-Lhoret R, McCrimmon RJ, Hume C, Annan F, Fournier PA, Graham C, Bode B, Galassetti P, Jones TW, Millan IS, Heise T, Peters AL, Petz A, Laffel LM. Exercise management in type 1 diabetes: a consensus statement. Lancet Diabetes Endocrinol. 2017 May;5(5):377-390. doi: 10.1016/S2213-8587(17)30014-1. Epub 2017 Jan 24. PMID 28126459
- [Background] Rogers MAM, Kim C, Banerjee T, Lee JM. Fluctuations in the incidence of type 1 diabetes in the United States from 2001 to 2015: a longitudinal study. BMC Med. 2017 Nov 8;15(1):199. doi: 10.1186/s12916-017-0958-6. PMID 29115947
- [Background] Watson JM, Jenkins EJ, Hamilton P, Lunt MJ, Kerr D. Influence of caffeine on the frequency and perception of hypoglycemia in free-living patients with type 1 diabetes. Diabetes Care. 2000 Apr;23(4):455-9. doi: 10.2337/diacare.23.4.455. PMID 10857934
- [Background] Silink M. Childhood diabetes: a global perspective. Horm Res. 2002;57 Suppl 1:1-5. doi: 10.1159/000053304. PMID 11979014
- [Background] Wysham C, Bhargava A, Chaykin L, de la Rosa R, Handelsman Y, Troelsen LN, Kvist K, Norwood P. Effect of Insulin Degludec vs Insulin Glargine U100 on Hypoglycemia in Patients With Type 2 Diabetes: The SWITCH 2 Randomized Clinical Trial. JAMA. 2017 Jul 4;318(1):45-56. doi: 10.1001/jama.2017.7117. PMID 28672317
- [Background] Zaharieva DP, Miadovnik LA, Rowan CP, Gumieniak RJ, Jamnik VK, Riddell MC. Effects of acute caffeine supplementation on reducing exercise-associated hypoglycaemia in individuals with Type 1 diabetes mellitus. Diabet Med. 2016 Apr;33(4):488-96. doi: 10.1111/dme.12857. Epub 2015 Aug 18. PMID 26173655
- [Background] Zaharieva DP, Riddell MC. Caffeine and glucose homeostasis during rest and exercise in diabetes mellitus. Appl Physiol Nutr Metab. 2013 Aug;38(8):813-22. doi: 10.1139/apnm-2012-0471. Epub 2013 May 14. PMID 23855268